CLINICAL TRIAL: NCT04093024
Title: A Double Blind, Randomised, Placebo-controlled Trial to Evaluate the Dose-exposure and Safety of Nintedanib Per os on Top of Standard of Care for 24 Weeks, Followed by Open Label Treatment With Nintedanib of Variable Duration, in Children and Adolescents (6 to 17 Year-old) With Clinically Significant Fibrosing Interstitial Lung Disease
Brief Title: A Study to Find Out How Nintedanib is Taken up in the Body and How Well it is Tolerated in Children and Adolescents With Interstitial Lung Disease (ILD)
Acronym: InPedILD®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199-0337; 2018-004530-14 (EudraCT Number)
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double-blind period (DBP) + open-label Nintedanib period (OLNP): Randomised Nintedanib (Experimental): This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP and OLNP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib in both periods (DBP + OLNP). Participants in this arm do not entail participants from the 'randomised to placebo' arms.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
  Interventions: Drug: Nintedanib
- DBP+OLNP: Randomised placebo (Placebo Comparator): Placebo randomised participants were treated orally with a Nintedanib matching placebo soft capsule twice daily in the double-blind period (DBP).
  Participants who continued with the open-label Nintedanib period (OLNP) after the DBP switched to active Nintedanib treatment in the OLNP and were treated orally with Nintedanib twice daily.
  Medication dosage was per administration 50 milligram (mg) [2 25 mg capsules (cap)],75 mg [3 25 mg cap], 100 mg [1 100 mg or 4 25 mg cap] or 150 mg [1 150 mg or 6 25 mg cap] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  The dose interval was approximately 12 hours between one and the next dose.
  Here participants received placebo first (DBP) and then Nintedanib (OLNP). DBP: Planned was from first to last randomised blinded drug intake. OLNP: Planned was from first to last open-label Nintedanib intake.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — Capsule
  Other Names: Ofev®
  Arms: Double-blind period (DBP) + open-label Nintedanib period (OLNP): Randomised Nintedanib
Drug: Placebo — Capsule
  Arms: DBP+OLNP: Randomised placebo

SUMMARY:
The main objective of the study is to evaluate dose-exposure and safety of nintedanib in children and adolescents with fibrosing Interstitial Lung Disease (ILD).

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents 6 to 17 years old at Visit 2.
* Signed and dated written informed consent and assent, where applicable, in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Male or female patients. Female of childbearing potential (WOCBP) must confirm that sexual abstinence is standard practice and will be continued until 3 months after last drug intake, or be ready and able to use a highly effective method of birth control per International Conference on Harmonisation (ICH) M3 (R2) that results in a low failure rate of less than 1% per year when used consistently and correctly, in combination with one barrier method, from 28 days prior to initiation of study treatment, during treatment and until 3 months after last drug intake. Sexual abstinence is defined as abstinence from any sexual act that may result in pregnancy. A list of contraception methods meeting these criteria is provided in the parental information.
* Patients with evidence of fibrosing Interstitial Lung Disease (ILD) on High-Resolution Computed Tomography (HRCT) within 12 months of Visit 1 as assessed by the investigator and confirmed by central review.
* Patients with Forced Vital Capacity (FVC)% predicted ≥25% at Visit 2. [Note: Predicted normal values will be calculated according to GLI (Global Lung Initiative)]
* Patients with clinically significant disease at Visit 2, as assessed by the investigator based on any of the following:

  * Fan score ≥3, or
  * Documented evidence of clinical progression over time based on either

    * a 5-10% relative decline in FVC% predicted accompanied by worsening symptoms, or
    * a ≥10% relative decline in FVC % predicted, or
    * increased fibrosis on HRCT, or
    * other measures of clinical worsening attributed to progressive lung disease (e.g. increased oxygen requirement, decreased diffusion capacity).

Exclusion Criteria:

* Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT)>1.5 x Upper Level of Normal (ULN) at Visit 1.
* Bilirubin >1.5 x ULN at Visit 1.
* Creatinine clearance <30 mL/min calculated by Schwartz formula at Visit 1. [Note: Laboratory parameters from Visit 1 have to satisfy the laboratory threshold values as shown above. Visit 2 laboratory results will be available only after randomization. In case at Visit 2 the results do no longer satisfy the entry criteria, the Investigator has to decide whether it is justified that the patient remains on study drug. The justification for decision needs to be documented. Laboratory parameters that are found to be abnormal at Visit 1 are allowed to be re-tested (once) if it is thought to be a measurement error (i.e. there was no abnormal result of this test in the recent history of the patient and there is no related clinical sign) or the result of a temporary and reversible medical condition, once that condition is resolved.]
* Patients with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment) at Visit 1.
* Previous treatment with nintedanib.
* Other investigational therapy received within 1 month or 5 half-lives (whichever is shorter but ≥1 week) prior to Visit 2.
* Significant pulmonary arterial hypertension (PAH) defined by any of the following:

  * Previous clinical or echocardiographic evidence of significant right heart failure
  * History of right heart catheterization showing a cardiac index ≤2 l/min/m²
  * PAH requiring parenteral therapy with epoprostenol/treprostinil
* In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
* Cardiovascular diseases, any of the following:

  * Severe hypertension, uncontrolled under treatment, within 6 months of Visit 1. Uncontrolled hypertension is defined as

    * In children 6 to ≤12 years old: ≥95th percentile + 12 mm Hg or ≥140/90 mm Hg (whichever is lower) (systolic or diastolic blood pressure equal to or greater than the calculated target value)
    * In adolescents 13 to 17 years old: systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg
  * Myocardial infarction within 6 months of Visit 1
  * Unstable cardiac angina within 6 months of Visit 1
* Bleeding risk, any of the following:

  * Known genetic predisposition to bleeding
  * Patients who require

    * Fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors, heparin, hirudin)
    * High dose antiplatelet therapy [Note: Prophylactic low dose heparin or heparin flush as needed for maintenance of an indwelling intravenous device (e.g. enoxaparin 4000 I.U. s.c. per day), as well as prophylactic use of antiplatelet therapy (e.g. acetyl salicylic acid up to 325 mg/day, or clopidogrel at 75 mg/day, or equivalent doses of other antiplatelet therapy) are not prohibited.]
  * History of haemorrhagic central nervous system (CNS) event within 12 months of Visit 1
  * Any of the following within 3 months of Visit 1:

    * Haemoptysis or haematuria
    * Active gastro-intestinal (GI) bleeding or GI - ulcers
    * Major injury or surgery (investigator's judgment)
  * Any of the following coagulation parameters at Visit 1:

    * International normalized ratio (INR) >2
    * Prolongation of prothrombin time (PT) by >1.5 x ULN
    * Prolongation of activated partial thromboplastin time (aPTT) by >1.5 x ULN
* History of thrombotic event (including stroke and transient ischemic attack) within 12 months of Visit 1.
* Known hypersensitivity to the trial medication or its components (i.e. soya lecithin).
* Patients with documented allergy to peanut or soya.
* Other disease that may interfere with testing procedures or in the judgment of the investigator may interfere with trial participation or may put the patient at risk when participating in this trial.
* Life expectancy for any concomitant disease other than Interstitial Lung Disease (ILD)<2.5 years (investigator assessment).
* Female patients who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Patients not able or willing to adhere to trial procedures, including intake of study medication.
* Patients with any diagnosed growth disorder such as growth hormone deficiency or any genetic disorder that is associated with short stature (e.g. Turner Syndrome, Noonan Syndrome, Russell-Silver Syndrome) and/or treatment with growth hormone therapy within 6 months before Visit 2. Patients with short stature considered by the investigator to be due to glucocorticoid therapy may be included.
* Patients <13.5 kg of weight at Visit 1 (same threshold to be used for male and female patients).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (9):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Weill Cornell Medicine, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seattle Children's Hospital, Seattle, Washington
- Argentina (3):
  - Hospital de Pediatría " Prof. Dr. Juan P. Garrahan", CABA
  - Hospital de Niños Dr. Ricardo Gutierrez, CABA
  - INSARES, Mendoza
- Women's and Children's Hospital, North Adelaide, South Australia, Australia
- Brussels - UNIV HUDERF, Brussels, Belgium
- Brazil (2):
  - Serviços Medicos Respirar Sul Fluminense, Barra Mansa
  - Centro de Pesquisa Clinica do Instituto da Crianca - HCFMUSP, São Paulo
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
- Teaching Hospital Motol, Oncology Clinic, Prague, Czechia
- Aarhus University Hospital, Aarhus N, Denmark
- Tampere University Hospital, Tampere, Finland
- France (2):
  - HOP Intercommunal, Créteil
  - HOP Armand-Trousseau, Paris
- General Hospital of Thessaloniki "Ippokrateio", Thessaloniki, Greece
- Semmelweis University, Budapest, Hungary
- Italy (3):
  - Azienda Ospedaliera Meyer, Florence
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Osp. Pediatrico Bambin Gesù, Roma
- Clinical Research Institute S.C., Tlalnepantla, Mexico
- Oslo Universitetssykehus HF, Rikshospitalet, Oslo, Norway
- Independent Public Teaching Children's Hospital, Warsaw, Poland
- Portugal (2):
  - CHULC, EPE - Hospital Dona Estefânia, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital Santa Maria, Lisbon
- Russia (3):
  - Children's Hematology,Oncology&Immunology na Rogachev,Moscow, Moscow
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - St. Petersburg State Pediatric University, Saint Petersburg
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Virgen del Rocío, Seville
- Ukraine (3):
  - Regional Children Clinical Hospital, Pulmonology, Kharkiv, Kharkiv
  - Institute of Phthisiology and Pulmonology n. a. F.G.Yanovsky, Kyiv
  - Regional clinical children hospital, Zaporizhya, Zaporizhya
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Deterding R, Young LR, DeBoer EM, Warburton D, Cunningham S, Schwerk N, Flaherty KR, Brown KK, Dumistracel M, Erhardt E, Bertulis J, Gahlemann M, Stowasser S, Griese M; InPedILD trial investigators. Nintedanib in children and adolescents with fibrosing interstitial lung diseases. Eur Respir J. 2023 Feb 2;61(2):2201512. doi: 10.1183/13993003.01512-2022. Print 2023 Feb. PMID 36041751
- [Derived] Deterding R, Griese M, Deutsch G, Warburton D, DeBoer EM, Cunningham S, Clement A, Schwerk N, Flaherty KR, Brown KK, Voss F, Schmid U, Schlenker-Herceg R, Verri D, Dumistracel M, Schiwek M, Stowasser S, Tetzlaff K, Clerisme-Beaty E, Young LR. Study design of a randomised, placebo-controlled trial of nintedanib in children and adolescents with fibrosing interstitial lung disease. ERJ Open Res. 2021 Jun 21;7(2):00805-2020. doi: 10.1183/23120541.00805-2020. eCollection 2021 Apr. PMID 34164554
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, multinational, prospective clinical trial to evaluate the dose-exposure and safety of Nintedanib on top of standard of care (SOC) in children and adolescents (6 to 17 years old) with clinically significant fibrosing Interstitial Lung Disease (ILD) in two parts. A randomised, placebo-controlled, double-blind treatment period of 24 weeks (double-blind period (DBP)) was followed by an open-label Nintedanib period (OLNP)) of variable duration.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All participants were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all participants was adhered to throughout the trial conduct. Treatment interruption and dose reduction were allowed as medically indicated.
Groups:
- DBP+OLNP: Randomised to Placebo: This arm shows placebo randomised participants treated orally with a Nintedanib matching placebo soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Participants who continued with the open-label Nintedanib period (OLNP) after the DBP switched to active Nintedanib treatment in the OLNP and were treated orally with Nintedanib twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received placebo first (DBP) and then Nintedanib (OLNP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
- DBP+OLNP: Randomised to Nintedanib: This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP and OLNP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib in both periods (DBP + OLNP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
Period: Double-blind Period
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Started | 13 | 26
Completed | 11 | 21
Not Completed | 2 | 5
Not completed — Completed prematurely due to administrative end of trial and did not continue with OLNP | 2 | 2
Not completed — Discontinued treatment due to adverse event | 0 | 2
Not completed — Discontinued treatment due to other reason | 0 | 1
Period: Open-label Nintedanib Period (OLNP)
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Started | 11 | 21
Completed | 11 | 20
Not Completed | 0 | 1
Not completed — Discontinuation of trial medication due to other reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS consisted of participants who were randomised to a treatment group and received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib | Total
Number analyzed (Participants) | 13 | 26 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.9 (2.8) | 12.5 (3.6) | 12.6 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 8 | 16 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 8 | 18 | 26
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 12 | 19 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve at Steady State (AUCτ,ss) Based on Sampling at Steady State (at Week 2 and Week 26)
Description: Area under the plasma concentration-time curve at steady state (AUCt,ss) based on sampling at steady state (at Week 2 and Week 26) after multiple oral administration of Nintedanib by age group over all treatments.
  Values of samples taken at Week 2 (for randomised Nintedanib participants) and at Week 26 (for randomised placebo participants) were used. Missing values at Week 2 of randomised Nintedanib participants were replaced with values taken at Week 26.
Time Frame: At Week 2 and at Week 26: at 5 minutes before and at 0, 1, 2, 3, 4, 6, and 8 hours post administration of the morning dose
Population: Pharmacokinetic parameter analysis set (PKS):
  This set includes all patients in the treated set (TS) who provide at least one pharmacokinetic (PK) endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours times nanogram per mililiter
Groups:
- DBP+OLNP: 6 to < 12 Years - Exposed to Nintedanib: This arm shows participants aged 6 to < 12 years old who were exposed to Nintedanib only, either randomised placebo (treated with Nintedanib in the OLNP only) and randomised Nintedanib (treated with Nintedanib in both, DBP and OLNP). The 6 to < 12 years old participant were treated orally with Nintedanib twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib only (OLNP or DBP+OLNP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
- DBP+OLNP: 12 to <18 Years - Exposed to Nintedanib: This arm shows participants aged 12 to <18 years old who were exposed to Nintedanib only either randomised placebo (treated with Nintedanib in the OLNP only) and randomised Nintedanib (treated with Nintedanib in both, DBP and OLNP). The 12 to 18 years old participant were treated orally with Nintedanib twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib only (OLNP or DBP+OLNP). Participants in this arm do not entail participants from the '6 to < 12 years - exposed to Nintedanib' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
Arm/Group | DBP+OLNP: 6 to < 12 Years - Exposed to Nintedanib | DBP+OLNP: 12 to <18 Years - Exposed to Nintedanib
Number analyzed (Participants) | 10 | 23
Hours times nanogram per mililiter | 175 (85.1) | 167 (83.6)

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events During the Double-blind Period
Description: Treatment-emergent was defined as: Adverse events with onset or worsening on or after date of treatment start until end of double-blind period (defined as the day before first intake of open-label nintedanib or last double-blind drug intake + residual effect period, whichever is earlier) were considered as treatment-emergent and were included in the analysis. Adverse events were counted under the treatment as randomized for the double-blind period.
Time Frame: From first drug administration until the earlier of (i) first intake of open-label nintedanib (exclusive) and (ii) last drug intake, up to 28 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- DBP: Randomised to Placebo: This arm shows placebo randomised participants treated orally with a Nintedanib matching placebo soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received placebo only (DBP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Nintedanib: This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Participants | 11 | 22

3. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Pathological Finding of Epiphyseal Growth Plate on Imaging up to Week 24, and Week 52
Description: Number of participants with at least one treatment-emergent pathological finding of the epiphyseal growth plate imaging (Magnetic Resonance Imaging (MRI)s/x-rays) were analyzed cumulatively and based on central review.
Time Frame: Up to Week 24 (included values at Week 12 and Week 24); Up to Week 52 (included values at Week 12, 24, 36 and 52)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Participants
  At Week 24 | 1 | 2
  At Week 52 | 2 | 3

4. Secondary Outcome: Number of Participants With Treatment-emergent Pathological Findings on Dental Examination or Imaging up to Week 24
Description: Number of participants with treatment-emergent pathological findings on dental examination (clinical examination) based on dentist assessment or imaging (panoramic x-ray) based on central review were analyzed. Number of participants with treatment-emergent pathological findings on dental imaging were analyzed cumulatively.
Time Frame: Dental examination: at Week 12 and Week 24; Dental imaging: at Week 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Participants
  Dental examination: Pathological findings up to week 24 | 1 | 5
  Dental imaging: Stunted growth of dental root | 0 | 6
  Dental imaging: Accelerated growth of dental root | 0 | 0
  Dental imaging: extra / supernumerary teeth | 0 | 0
  Dental imaging: Impacted permanent teeth | 2 | 4
  Dental imaging: Additional findings | 1 | 5
  Dental imaging: Other findings | 2 | 1

5. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Pathological Findings on Dental Examination or Imaging up to Week 52
Description: as for outcome 4
Time Frame: Dental examination: at Week 12, 24, 34, and Week 52; Dental imaging: at Week 24 and at Week 52.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Participants
  Dental examination: Pathological findings up to week 52 | 3 | 7
  Dental imaging: Stunted growth of dental root | 0 | 6
  Dental imaging: Accelerated growth of dental root | 0 | 0
  Dental imaging: extra / supernumerary teeth | 0 | 0
  Dental imaging: Impacted permanent teeth | 2 | 5
  Dental imaging: Additional findings | 1 | 6
  Dental imaging: Other findings | 3 | 2

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Over the Whole Trial
Description: Treatment-emergent was defined as: Adverse events with onset or worsening on or after date of treatment start until last drug intake + residual effect period was considered as treatment-emergent and was included in the analysis. Adverse events were counted under the treatment as randomized for the double-blind period.
Time Frame: From first drug administration until the last drug intake, up to 92 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- DBP: Randomised to Placebo: This arm shows placebo randomised participants treated orally with a Nintedanib matching soft capsules twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP) up to week 24.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received placebo only (DBP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- OLNP: Randomised to Placebo and Switched to Nintedanib: This arm shows participants who continued with the open-label Nintedanib period (OLNP) after the DBP, switched to active Nintedanib treatment in the OLNP and were treated orally with Nintedanib twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib only (OLNP).
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
- DBP+OLNP: Randomised to Nintedanib: This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP and OLNP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib in both periods (DBP + OLNP). Participants in this arm do not entail participants from the 'randomised to placebo' arms.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
Arm/Group | DBP: Randomised to Placebo | OLNP: Randomised to Placebo and Switched to Nintedanib | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 11 | 26
Participants | 11 | 11 | 26

7. Secondary Outcome: Absolute Change From Baseline in Height at Week 24
Description: Absolute change from baseline in height at Week 24 was measured with a stadiometer 3 times at each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in height at Week 24 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: MMRM included measurements pre-administration at -4 weeks and at 0, 12, 24, 36, 52, 64, 76, and 88 weeks after first drug administration. MMRM values at Week 24 are reported in the table below
Population: Treated set (TS): The TS consisted of participants who were randomised to a treatment group and received at least one dose of study medication. Only participants with correctly measured baseline and at least one post-baseline measurement were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeter
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 25
Centimeter | 1.3 [0.6 to 1.9] | 1.3 [0.8 to 1.8]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; No formal hypotheses were tested; Test type: Other; p = 0.9858, Mixed Model Repeated Measures (MMRM); Fixed categorical effects: (Randomised) treatment, age-group; Fixed continuous effects: Baseline at each visit, random effect for participant; Adjusted mean difference = 0.0, 95% CI 2-sided [-0.8 to 0.8], Standard Error of Mean 0.4 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

8. Secondary Outcome: Absolute Change From Baseline in Height at Week 52
Description: Absolute change from baseline in height at Week 52 was measured with a stadiometer 3 times at each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in height at Week 52 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: MMRM included measurements pre-administration at -4 weeks and at 0, 12, 24, 36, 52, 64, 76, and 88 weeks after first drug administration. MMRM values at Week 52 are reported in the table below
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeter
Groups:
- DBP+OLNP: Randomised to Nintedanib: This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP and OLNP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 25
Centimeter | 2.8 [1.5 to 4.2] | 2.8 [1.8 to 3.8]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised to Nintedanib; No formal hypotheses were tested; Test type: Other; p = 0.9769, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted mean difference = -0.0, 95% CI 2-sided [-1.7 to 1.6], Standard Error of Mean 0.8 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

9. Secondary Outcome: Absolute Change From Baseline in Height at Week 76
Description: Absolute change from baseline in height at Week 76 was measured with a stadiometer 3 times at each time point. The average of these 3 measurements was taken per time point.
  MMRM has been calculated but did not provide estimates for this time point due to low sample size. Thus, change in height from baseline to Week 76 was analyzed descriptively only.
Time Frame: Measurements were assessed at Week 0 and at Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 3 | 4
Centimeter
  At Baseline | 143.7 (11.2) | 162.5 (15.8)
  At Week 76 | 150.0 (15.7) | 165.5 (13.0)

10. Secondary Outcome: Absolute Change From Baseline in Sitting Height at Week 24
Description: Absolute change from baseline in sitting height at Week 24 was measured with a stadiometer 3 times at each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in sitting height at Week 24 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeters
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 6 | 15
Centimeters | 1.0 [-1.3 to 3.4] | 2.1 [0.6 to 3.6]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.4442, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 1.1, 95% CI 2-sided [-1.8 to 4.0], Standard Error of Mean 1.4 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

11. Secondary Outcome: Absolute Change From Baseline in Sitting Height at Week 52
Description: Absolute change from baseline in sitting height at Week 52 was measured with a stadiometer 3 times at each time point. The average of these 3 measurements was taken per time point.
  MMRM has been calculated but did not provide estimates for this time point due to low sample size. Thus, change in sitting height from baseline to Week 52 was analyzed descriptively only.
Time Frame: Measurements were assessed at Week 0 and at Week 52
Population: Treated set (TS): The TS consisted of participants who were randomised to a treatment group and received at least one dose of study medication. Only participants with non-missing results were included in the analysis.
Measure: Mean (Standard Deviation); unit: Centimeters
Groups:
- DBP + OLNP: Randomised to Placebo: This arm shows placebo randomised participants treated orally with a Nintedanib matching placebo soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Participants who continued with the open-label Nintedanib period (OLNP) after the DBP switched to active Nintedanib treatment in the OLNP and were treated orally with Nintedanib twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received placebo first (DBP) and then Nintedanib (OLNP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
- DBP + OLNP: Randomised to Nintedanib: This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP and OLNP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib in both periods (DBP + OLNP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
Arm/Group | DBP + OLNP: Randomised to Placebo | DBP + OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 3 | 7
Centimeters
  At Baseline | 78.7 (11.8) | 77.6 (9.4)
  At Week 52 | 79.0 (12.2) | 79.3 (8.6)

12. Secondary Outcome: Absolute Change From Baseline in Sitting Height at Week 76
Description: Absolute change from baseline in sitting height at Week 76 was measured with a stadiometer 3 times at each time point. The average of these 3 measurements was take per time point.
  MMRM has been calculated but did not provide estimates for this time point due to low sample size. Thus, change in sitting height from baseline to Week 76 was analyzed descriptively only.
Time Frame: Measurements were assessed at Week 0 and at Week 76
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | DBP + OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 1 | 2
Centimeters
  At Baseline | 65.0 (NA) — One participant is not sufficient to calculate a standard deviation. | 83.0 (4.2)
  At Week 76 | 65.0 (NA) — One participant is not sufficient to calculate a standard deviation. | 84.5 (3.5)

13. Secondary Outcome: Absolute Change From Baseline in Leg Length at Week 24 - Left
Description: Absolute change from baseline in left leg length at Week 24 was assessed by measuring the distance between the anterior iliac spine and the medial malleolus 3 times at each leg and each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in left leg length at Week 24 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: MMRM included measurements at 0, 12, 24, 36, 52, 64, and 76 weeks after first drug administration. MMRM values at Week 24 are reported in the table below
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeters
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 23
Centimeters | 1.6 [0.3 to 2.9] | 1.7 [0.8 to 2.7]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.8820, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 0.1, 95% CI 2-sided [-1.5 to 1.8], Standard Error of Mean 0.8 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

14. Secondary Outcome: Absolute Change From Baseline in Leg Length at Week 52 - Left
Description: Absolute change from baseline in left leg length at Week 52 was assessed by measuring the distance between the anterior iliac spine and the medial malleolus 3 times at each leg and each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in left leg length at Week 52 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: MMRM included measurements at 0, 12, 24, 36, 52, 64, and 76 weeks after first drug administration. MMRM values at Week 52 are reported in the table below
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeter
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 23
Centimeter | 2.8 [0.3 to 5.4] | 2.9 [0.9 to 4.9]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised to Nintedanib; No formal hypotheses were tested; Test type: Other; p = 0.9652, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted mean difference = 0.1, 95% CI 2-sided [-3.2 to 3.3], Standard Error of Mean 1.6 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

15. Secondary Outcome: Absolute Change From Baseline in Leg Length at Week 76 - Left
Description: Absolute change from baseline in left leg length at Week 76 was assessed by measuring the distance between the anterior iliac spine and the medial malleolus 3 times at each leg and each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in left leg length at Week 76 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: MMRM included measurements at 0, 12, 24, 36, 52, 64, and 76 weeks after first drug administration. MMRM values at Week 76 are reported in the table below
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeter
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 23
Centimeter | 5.2 [-0.0 to 10.5] | 2.6 [-1.5 to 6.7]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised to Nintedanib; No formal hypotheses were tested; Test type: Other; p = 0.4084, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted mean difference = -2.6, 95% CI 2-sided [-9.3 to 4.0], Standard Error of Mean 3.1 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

16. Secondary Outcome: Absolute Change From Baseline in Leg Length at Week 24 - Right
Description: Absolute change from baseline in right leg length at Week 24 was assessed by measuring the distance between the anterior iliac spine and the medial malleolus 3 times at each leg and each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in right leg length at Week 24 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 13
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeters
Groups:
- DBP: Randomised to Nintedanib: This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arms.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 23
Centimeters | 1.6 [0.3 to 2.9] | 1.6 [0.6 to 2.6]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.9928, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 0.0, 95% CI 2-sided [-1.6 to 1.6], Standard Error of Mean 0.8 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

17. Secondary Outcome: Absolute Change From Baseline in Leg Length at Week 52 - Right
Description: Absolute change from baseline in right leg length at Week 52 was assessed by measuring the distance between the anterior iliac spine and the medial malleolus 3 times at each leg and each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in right leg length at Week 52 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 14
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeter
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 23
Centimeter | 2.8 [0.4 to 5.1] | 3.4 [1.6 to 5.2]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised to Nintedanib; No formal hypotheses were tested; Test type: Other; p = 0.6366, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted mean difference = 0.7, 95% CI 2-sided [-2.3 to 3.6], Standard Error of Mean 1.4 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

18. Secondary Outcome: Absolute Change From Baseline in Leg Length at Week 76 - Right
Description: Absolute change from baseline in right leg length at Week 76 was assessed by measuring the distance between the anterior iliac spine and the medial malleolus 3 times at each leg and each time point. The average of these 3 measurements was taken per time point.
  Absolute change from baseline in right leg length at Week 76 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 15
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Centimeter
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 23
Centimeter | 3.9 [-0.5 to 8.3] | 4.3 [0.8 to 7.7]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised to Nintedanib; No formal hypotheses were tested; Test type: Other; p = 0.8823, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted mean difference = 0.4, 95% CI 2-sided [-5.2 to 5.9], Standard Error of Mean 2.3 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

19. Secondary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC) % Predicted at Week 24
Description: Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. The predicted values were calculated according to the Global Lungs Initiative (GLI) 2012 equations.
  Absolute change from baseline in Forced Vital Capacity (FVC) % predicted at Week 24 in the treated set(TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: MMRM included measurements pre-administration at -4 weeks and at 0, 2, 6, 12, 24, 26, 36, and 52 weeks after first drug administration. MMRM values at Week 24 are reported in the table below
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of predicted FVC
Groups:
- DBP: Randomised to Nintedanib: This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP and OLNP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Percentage of predicted FVC | -0.8939 [-4.6090 to 2.8211] | 0.3112 [-2.3595 to 2.9820]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.5962, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 1.2052, 95% CI 2-sided [-3.3966 to 5.8070], Standard Error of Mean 2.2491 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

20. Secondary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC) % Predicted at Week 52
Description: Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. The predicted values were calculated according to the Global Lungs Initiative (GLI) 2012 equations.
  Absolute change from baseline in Forced Vital Capacity (FVC) % predicted at Week 52 in the treated set(TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: MMRM included measurements pre-administration at -4 weeks and at 0, 2, 6, 12, 24, 26, 36, and 52 weeks after first drug administration. MMRM values at Week 52 are reported in the table below
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of predicted FVC
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP + OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Percentage of predicted FVC | -0.9827 [-6.2611 to 4.2958] | 0.7906 [-2.9464 to 4.5277]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP + OLNP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.5776, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 1.7733, 95% CI 2-sided [-4.7015 to 8.2481], Standard Error of Mean 3.1424 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

21. Secondary Outcome: Absolute Change From Baseline in Pediatric Quality of Life Questionnaire™(PedsQL™) at Week 24 - Parent Report
Description: The PedsQL™ questionnaires consists of 23 items (i) and 4 dimensions: physical (8i), emotional (5i), social (5i) and school (5i) functioning. A 5-point Likert response scale (0 = never (worst outcome) to 4=almost always (best outcome)) was used except for the Young Child Report, where a 3-point scale (0=not at all (worst outcome) to 4=a lot (best outcome)) was used. Items were reverse-scored and linearly transformed to a 0-100 scale (0 = 100 to 4 = 0). Higher scores indicated better health-related quality of life. To create total scores, the mean was computed.
  Absolute change from baseline in PedsQL™ reported by parents was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: MMRM included measurements at 0, 24, and 52 weeks after first drug administration. MMRM values at Week 24 are reported in the table below
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 11 | 21
Unit on scale | 5.615 [-1.506 to 12.736] | 5.481 [0.384 to 10.578]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.9755, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = -0.134, 95% CI 2-sided [-8.975 to 8.707], Standard Error of Mean 4.316 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

22. Secondary Outcome: Absolute Change From Baseline in Pediatric Quality of Life Questionnaire™(PedsQL™) at Week 52 - Parent Report
Description: as for outcome 21
Time Frame: MMRM included measurements at 0, 24, and 52 weeks after first drug administration. MMRM values at Week 52 are reported in the table below
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 11 | 21
Unit on scale | 4.377 [-4.403 to 13.157] | 7.830 [1.799 to 13.862]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.5140, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 3.453, 95% CI 2-sided [-7.250 to 14.157], Standard Error of Mean 5.225 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

23. Secondary Outcome: Absolute Change From Baseline in Pediatric Quality of Life Questionnaire™(PedsQL™) at Week 24 - Participant Report
Description: The PedsQL™ questionnaires consists of 23 items (i) and 4 dimensions: physical (8i), emotional (5i), social (5i) and school (5i) functioning. A 5-point Likert response scale (0 = never (worst outcome) to 4=almost always (best outcome)) was used except for the Young Child Report, where a 3-point scale (0=not at all (worst outcome) to 4=a lot (best outcome)) was used. Items were reverse-scored and linearly transformed to a 0-100 scale (0 = 100 to 4 = 0). Higher scores indicated better health-related quality of life. To create total scores, the mean was computed.
  Absolute change from baseline in PedsQL™ was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 11 | 21
Unit on scale | 5.484 [-0.051 to 11.018] | 6.514 [2.531 to 10.497]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.7613, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 1.030, 95% CI 2-sided [-5.848 to 7.908], Standard Error of Mean 3.358 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

24. Secondary Outcome: Absolute Change From Baseline in Pediatric Quality of Life Questionnaire™(PedsQL™) at Week 52 - Participant Report
Description: as for outcome 23
Time Frame: as for outcome 22
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 11 | 21
Unit on scale | 0.902 [-7.616 to 9.420] | 1.243 [-4.598 to 7.083]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.9468, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 0.340, 95% CI 2-sided [-10.026 to 10.707], Standard Error of Mean 5.049 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

25. Secondary Outcome: Absolute Change From Baseline in Oxygen Saturation (SpO₂) on Room Air at Rest at Week 24
Description: Oxygen saturation (SpO₂) was measured after minimum 5 minutes on room air by standard pulse oximetry at rest.
  Absolute change from baseline in SpO₂ at Week 24 in the treated set(TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 19
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of SpO₂
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Percentage of SpO₂ | -2.25 [-4.45 to -0.04] | 0.07 [-1.49 to 1.63]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.0908, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 2.31, 95% CI 2-sided [-0.39 to 5.02], Standard Error of Mean 1.33 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

26. Secondary Outcome: Absolute Change From Baseline in Oxygen Saturation (SpO₂) on Room Air at Rest at Week 52
Description: Oxygen saturation (SpO₂) was measured after minimum 5 minutes on room air by standard pulse oximetry at rest.
  Absolute change from baseline in SpO₂ at Week 52 in the treated set(TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 20
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of SpO₂
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Percentage of SpO₂ | -2.60 [-5.02 to -0.18] | -0.32 [-2.03 to 1.40]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.1222, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 2.28, 95% CI 2-sided [-0.69 to 5.25], Standard Error of Mean 1.39 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

27. Secondary Outcome: Absolute Change From Baseline in 6 Minutes (Min) Walk Distance at Week 24
Description: Absolute change from baseline in 6 minutes (min) walk distance at Week 24 in the treated set (TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Meter
Arm/Group | DBP: Randomised to Placebo | DBP: Randomised to Nintedanib
Number analyzed (Participants) | 11 | 21
Meter | 10.5 [-36.4 to 57.3] | 17.6 [-16.2 to 51.5]
Statistical Analysis 1: Comparison: DBP: Randomised to Placebo vs DBP: Randomised to Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.8012, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = 7.2, 95% CI 2-sided [-50.7 to 65.0], Standard Error of Mean 28.2 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

28. Secondary Outcome: Absolute Change From Baseline in 6 Minutes (Min) Walk Distance at Week 52
Description: Absolute change from baseline in 6 minutes (min) walk distance at Week 52 in the treated set(TS) was based on a Mixed Model Repeated Measures (MMRM), with fixed categorical effects of (randomised) treatment at each visit, age-group and the fixed continuous effects of baseline at each visit, and random effect for participant. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-participant measurements.
Time Frame: as for outcome 22
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Meter (m)
Groups:
- DBP+OLNP: Randomised Nintedanib: This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP and OLNP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib in both periods (DBP + OLNP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake, up to 24 weeks.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised Nintedanib
Number analyzed (Participants) | 11 | 21
Meter (m) | 28.1 [-29.4 to 85.5] | -4.9 [-44.5 to 34.7]
Statistical Analysis 1: Comparison: DBP+OLNP: Randomised to Placebo vs DBP+OLNP: Randomised Nintedanib; Test type: Other — No formal hypotheses were tested; p = 0.3401, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 7, analysis 1]; Adjusted Mean Difference = -32.9, 95% CI 2-sided [-103.1 to 37.2], Standard Error of Mean 33.8 — Adjusted mean difference was calculated as 'Randomised Nintedanib - randomised placebo'

29. Secondary Outcome: Participants Acceptability Based on the Size of Capsules at Week 24 - Patient Question
Description: Acceptability is defined as the overall ability and willingness of the participant to use the medicinal product as intended.
  Acceptability based on the capsule size was assessed by a acceptability questionnaire (1 item with 3 categories as shown below) for participants. In case the participant was considered not old enough as per investigator judgment the caregiver could assist with the completion.
  In addition to the commercially available 100 milligram (mg) soft capsules (oblong shape, 6 millimeter (mm) diameter and 16 mm length) and 150 mg soft capsules (oblong shape, 7 mm diameter and 18 mm length), 25 mg Nintedanib soft capsules of smaller size (oval shape, 5 mm diameter and 8 mm length) were provided in this trial for participants who were assigned to a dose smaller than 100 mg or were unable to swallow the larger 100 mg or 150 mg capsules.
Time Frame: Acceptability was assessed at Week 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- DBP: Randomised to Placebo - Capsule Size of 25 mg Capsule: This arm shows placebo randomised participants treated orally with placebo soft capsules of 25 milligram (mg) with a capsule size of 5 millimeter (mm) diameter and 8 mm length, oval shaped, twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage per administration was 50 milligram (mg) [2 capsules with strength 25 mg], 75 mg [3 capsules with strength 25 mg], 100 mg [4 capsules with strength 25 mg] or 150 mg [6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received placebo only (DBP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Nintedanib - Capsule Size of 25 mg Capsule: This arm shows Nintedanib randomised participants treated orally with Nintedanib soft capsules of 25 milligram (mg) with a capsule size of 5 millimeter (mm) diameter and 8 mm length, oval shaped, twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage per administration was 50 milligram (mg) [2 capsules with strength 25 mg], 75 mg [3 capsules with strength 25 mg], 100 mg [4 capsules with strength 25 mg] or 150 mg [6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Placebo - Capsule Size of 100 mg Capsule: This arm shows placebo randomised participants treated orally with placebo soft capsules of 100 mg with a capsule size of 6 mm diameter and 16 mm length, oblong shaped, twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage per administration was 100 mg [1 capsules with strength 100 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received placebo only (DBP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Nintedanib - Capsule Size of 100 mg Capsule: This arm shows Nintedanib randomised participants treated orally with Nintedanib soft capsules of 100 mg with a capsule size of 6 mm diameter and 16 mm length, oblong shaped, twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage per administration was 100 mg [1 capsules with strength 100 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Placebo - Capsule Size of 150 mg Capsule: This arm shows placebo randomised participants treated orally with placebo soft capsules of 150 mg with a capsule size of 7 mm diameter and 18 mm length, oblong shaped, twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage per administration was 150 mg [1 capsules with strength 150 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received placebo only (DBP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Nintedanib - Capsule Size of 150 mg Capsule: This arm shows Nintedanib randomised participants treated orally with Nintedanib soft capsules of 150 mg with a capsule size of 7 mm diameter and 18 mm length, oblong shaped, twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage per administration was 150 mg [1 capsules with strength 150 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
Arm/Group | DBP: Randomised to Placebo - Capsule Size of 25 mg Capsule | DBP: Randomised to Nintedanib - Capsule Size of 25 mg Capsule | DBP: Randomised to Placebo - Capsule Size of 100 mg Capsule | DBP: Randomised to Nintedanib - Capsule Size of 100 mg Capsule | DBP: Randomised to Placebo - Capsule Size of 150 mg Capsule | DBP: Randomised to Nintedanib - Capsule Size of 150 mg Capsule
Number analyzed (Participants) | 4 | 6 | 4 | 14 | 3 | 2
Participants
  OK | 4 | 6 | 4 | 14 | 3 | 2
  Large | 0 | 0 | 0 | 0 | 0 | 0
  Very Large | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Participants Acceptability Based on the Size of Capsules at Week 24 - Investigator Question
Description: Acceptability is defined as the overall ability and willingness of the participant to use the medicinal product as intended.
  Acceptability based on the capsule size was assessed by a acceptability questionnaire (1 item with 3 categories as shown below) for investigators.
  In addition to the commercially available 100 milligram (mg) soft capsules (oblong shape, 6 millimeter (mm) diameter and 16 mm length) and 150 mg soft capsules (oblong shape, 7 mm diameter and 18 mm length), 25 mg Nintedanib soft capsules of smaller size (oval shape, 5 mm diameter and 8 mm length) were provided in this trial for participants who were assigned to a dose smaller than 100 mg or were unable to swallow the larger 100 mg or 150 mg capsules.
Time Frame: Acceptability was assessed at Week 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DBP: Randomised to Placebo - Capsule Size of 25 mg Capsule | DBP: Randomised to Nintedanib - Capsule Size of 25 mg Capsule | DBP: Randomised to Placebo - Capsule Size of 100 mg Capsule | DBP: Randomised to Nintedanib - Capsule Size of 100 mg Capsule | DBP: Randomised to Placebo - Capsule Size of 150 mg Capsule | DBP: Randomised to Nintedanib - Capsule Size of 150 mg Capsule
Number analyzed (Participants) | 4 | 6 | 4 | 14 | 3 | 2
Participants
  No | 1 | 2 | 1 | 2 | 0 | 1
  Yes | 0 | 0 | 0 | 0 | 0 | 0
  Missing | 3 | 4 | 3 | 12 | 3 | 1

31. Secondary Outcome: Participants Acceptability Based on the Number of Capsules at Week 24 - Patient Question
Description: Acceptability is defined as the overall ability and willingness of the participant to use the medicinal product as intended.
  Acceptability based on the number of capsule was assessed by a acceptability questionnaire (1 item with 3 categories as shown below) for participants. In case the participant was considered not old enough as per investigator judgment the caregiver could assist with the completion.
  In addition to the commercially available 100 milligram (mg) soft capsules (oblong shape, 6 millimeter (mm) diameter and 16 mm length) and 150 mg soft capsules (oblong shape, 7 mm diameter and 18 mm length), 25 mg Nintedanib soft capsules of smaller size (oval shape, 5 mm diameter and 8 mm length) were provided in this trial for participants who were assigned to a dose smaller than 100 mg or were unable to swallow the larger 100 mg or 150 mg capsules. Medication dosage was based on the participant's body weight and number of capsules per administration ranged from 2 to >6 capsules.
Time Frame: Acceptability was assessed at Week 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- DBP: Randomised to Placebo - 2 Capsules: This arm shows placebo randomised participants treated orally with 1 Nintedanib matching placebo soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 100 mg [1 capsule with strength 100 mg] or 150 mg [1 capsule with strength 150 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received placebo only (DBP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Nintedanib - 2 Capsules: This arm shows Nintedanib randomised participants treated orally with 1 Nintedanib soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 100 mg [1 capsule with strength 100 mg] or 150 mg [1 capsule with strength 150 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Placebo - 4 Capsules: This arm shows placebo randomised participants treated orally with 2 Nintedanib matching placebo soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg], based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received placebo only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Nintedanib - 4 Capsules: This arm shows Nintedanib randomised participants treated orally with 2 Nintedanib soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg], based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Placebo - 6 Capsules: This arm shows placebo randomised participants treated orally with 3 Nintedanib matching placebo soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 75 mg [3 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received placebo only (DBP).
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Nintedanib - 6 Capsules: This arm shows Nintedanib randomised participants treated orally with 3 Nintedanib soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 75 mg [3 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Placebo - >6 Capsules: This arm shows placebo randomised participants treated orally with >3 Nintedanib matching placebo soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 100 mg [4 capsules with strength 25 mg] or 150 mg [6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received placebo only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
- DBP: Randomised to Nintedanib - >6 Capsules: This arm shows Nintedanib randomised participants treated orally with >3 Nintedanib soft capsule twice daily with a dose interval of approximately 12 hours from one dose to the next dose in the double-blind period (DBP).
  Medication dosage was per administration 100 mg [4 capsules with strength 25 mg] or 150 mg [6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks).
  In this arm participants received Nintedanib only (DBP). Participants in this arm do not entail participants from the 'randomised to placebo' arm.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
Arm/Group | DBP: Randomised to Placebo - 2 Capsules | DBP: Randomised to Nintedanib - 2 Capsules | DBP: Randomised to Placebo - 4 Capsules | DBP: Randomised to Nintedanib - 4 Capsules | DBP: Randomised to Placebo - 6 Capsules | DBP: Randomised to Nintedanib - 6 Capsules | DBP: Randomised to Placebo - >6 Capsules | DBP: Randomised to Nintedanib - >6 Capsules
Number analyzed (Participants) | 7 | 16 | 2 | 3 | 1 | 3 | 1 | 0
Participants
  I had no problem swallowing them | 7 | 16 | 2 | 3 | 1 | 3 | 1 | 0
  I swallowed them but it was difficult | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  I could not swallow them sometimes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Number of Participants With Occurrence of First Respiratory-related Hospitalization Over the Whole Trial
Description: Number of participants with occurrence of first respiratory-related hospitalization over the whole trial.
  The number of participants with first respiratory-related hospitalization is reported instead of a metric summarizing the time-to-event data with unit of time, as the numbers resulting from the Kaplan-Meier-analysis were even below the first quartile.
Time Frame: From first drug administration until the last drug intake + 28 days residual effect period (REP), up to 92.6 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Participants | 0 | 3

33. Secondary Outcome: Number of Participants With Occurrence of First Acute Interstitial Lung Disease (ILD) Exacerbation or Death Over the Whole Trial
Description: Number of participants with occurrence of first acute Interstitial Lung Disease (ILD) exacerbation or death over the whole trial. The number of participants with first acute ILD exacerbation is reported instead of a metric summarizing the time-to-event data with unit of time, as the numbers resulting from the Kaplan-Meier-analysis were even below the first quartile.
Time Frame: From first drug administration until the last drug intake + 28 days REP, up to 92.6 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Participants | 0 | 2

34. Secondary Outcome: Number of Participants With Occurrence of Death Over the Whole Trial
Description: Number of participants with occurrence of death over the whole trial over the whole trial was computed. The number of participants with occurrence of death is reported instead of a metric summarizing the time-to-event data with unit of time, as the numbers resulting from the Kaplan-Meier-analysis were even below the first quartile.
Time Frame: From first drug administration until the last drug intake + 28 days REP, up to 92.6 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DBP+OLNP: Randomised to Placebo | DBP+OLNP: Randomised to Nintedanib
Number analyzed (Participants) | 13 | 26
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Placebo-randomised DBP: From treatment start till end of DBP (defined as the day before first intake of open-label nintedanib (NIN) or last double-blind drug intake, up to 24.4 weeks + 28 days (REP), whichever is earlier) Placebo-randomised OLNP: From first intake of NIN till last intake of the OLNP, up to 64.6 weeks + 28 days (REP). Nintedanib-randomised DBP+OLNP: From first intake of NIN (DBP / OLNP) till last intake of NIN (DBP or OLNP), up to 85.1 weeks + 28 days (REP).
Description: Treated set (TS): The TS consisted of participants who were randomised to a treatment group and received at least one dose of study medication.
Groups:
- DBP+OLNP: Randomised to Nintedanib (Nintedanib Exposure Period): This arm shows Nintedanib randomised participants treated orally with Nintedanib in the DBP and OLNP twice daily with a dose interval of approximately 12 hours from one dose to the next dose.
  Medication dosage was per administration 50 milligram (mg) [2 capsules with strength 25 mg],75 mg [3 capsules with strength 25 mg], 100 mg [1 capsule with strength 100 mg or 4 capsules with strength 25 mg] or 150 mg [1 capsule with strength 150 mg or 6 capsules with strength 25 mg] based on the participant's weight at baseline (= 0 weeks). The dosage was adjusted at subsequent visits if the participant's weight had changed.
  In this arm participants received Nintedanib in both periods (DBP + OLNP). Participation in this arm do not entail participants from the 'randomised to placebo' arms.
  DBP: Planned was from first randomised trial drug intake to last blinded drug intake.
  OLNP: Planned was from first open-label Nintedanib intake to last open-label Nintedanib intake.
Arm/Group | DBP: Randomised to Placebo | OLNP: Randomised to Placebo and Switched to Nintedanib | DBP+OLNP: Randomised to Nintedanib (Nintedanib Exposure Period)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/13 | 2/11 | 5/26
Other Adverse Events (participants affected / at risk) | 11/13 | 11/11 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBP: Randomised to Placebo (N=13) | OLNP: Randomised to Placebo and Switched to Nintedanib (N=11) | DBP+OLNP: Randomised to Nintedanib (Nintedanib Exposure Period) (N=26)
Tooth development disorder (Gastrointestinal disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 2
Carbon dioxide increased (Investigations) | 0 | 0 | 1
Frontal lobe epilepsy (Nervous system disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Neurogenic shock (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DBP: Randomised to Placebo (N=13) | OLNP: Randomised to Placebo and Switched to Nintedanib (N=11) | DBP+OLNP: Randomised to Nintedanib (Nintedanib Exposure Period) (N=26)
Right atrial hypertrophy (Cardiac disorders) | 0 | 1 | 0
Supernumerary teeth (Congenital, familial and genetic disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Dental caries (Gastrointestinal disorders) | 3 | 1 | 7
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 12
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 2 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Malpositioned teeth (Gastrointestinal disorders) | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 6 | 6
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Tooth deposit (Gastrointestinal disorders) | 0 | 1 | 0
Tooth development disorder (Gastrointestinal disorders) | 1 | 0 | 6
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 4 | 7
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 2
Fatigue (General disorders) | 2 | 0 | 2
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 4
Multiple allergies (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 7
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 2
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 2
SARS-CoV-2 test positive (Investigations) | 0 | 2 | 1
Weight decreased (Investigations) | 0 | 0 | 2
X-ray limb abnormal (Investigations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 3
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Bruxism (Psychiatric disorders) | 0 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Melanosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
In the protocol it was planned to communicate the end of trial (EoT) once 30 participants had completed pharmacokinetic (PK) sampling at Week 26 or prematurely discontinued the trial and PK data was confirmed as adequate.

When the EoT was communicated, no participant had reached Week 100 yet, thus Week 100 time points were not assessable and the trial was completed as per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT04093024/Prot_002.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04093024/SAP_001.pdf